CLINICAL TRIAL: NCT05251623
Title: The Effect of Walking Program With Pedometer on Quality-of-life Among Chronic Obstructive Pulmonary Disease Patients
Brief Title: Walking Program With Pedometer on Quality of Life in COPD
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Chen Yen-Huey, assist professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TYGH106081
Record Dates: First submitted 2021-12-30; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; pedometer; physical activity; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pedometer (Experimental): walking with pedometer
  Interventions: Other: walking program
- control (No Intervention): no intervention

INTERVENTIONS:
Other: walking program — Subjects in PG walked to target steps daily with pedometer for 6 weeks
  Arms: pedometer

SUMMARY:
The aim of this study is to investigate the effects of a walking program on exercise capacity and quality of life in patient with COPD. Method: Patients with COPD were randomly assigned to pedometer group (PG) or control group (CON). Subjects in PG walked to target steps daily with pedometer for 6 weeks. Before and after the program, the following measurements were performed: pulmonary function test (PFT), daily steps, Six-Minute Walk Test (6MWT), COPD Assessment Test (CAT), and quality of life questionnaire (SF-12).

DETAILED DESCRIPTION:
Patients with chronic obstructive pulmonary disease (COPD) are suffered from impaired pulmonary function and dyspnea which result to limited level of physical activity, and impaired quality of life. Exercise and regular physical activity have been proven to break the vicious circle. The aim of this study is to investigate the effects of a walking program on exercise capacity and quality of life in patient with COPD. Method: Patients with COPD were randomly assigned to pedometer group (PG) or control group (CON). Subjects in PG walked to target steps daily with pedometer for 6 weeks. Before and after the program, the pulmonary function was assessed by spiromtery test. The exercise capacity were assessed by six-minute walking test, the physical activity level was assessed by daily steps, The quality of life was assessed by COPD Assessment Test (CAT), and quality of life questionnaire (SF-12).

.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with COPD
2. in a medically stable condition
3. able to walk unassisted
4. ≥ 40 years of age

Exclusion Criteria:

1. oxygen therapy,
2. hemodynamic instability,
3. signs/symptoms of acute infection
4. severe neurological, musculoskeletal, or cardiovascular conditions that affect walking

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
tidal volume | week 0
  the amount of air that moves in or out of the lungs with each respiratory cycle. It is measured by spirometers.
tidal volume | week 7
  the amount of air that moves in or out of the lungs with each respiratory cycle. It is measured by spirometers.
Short-form 12 questionnaire (SF-12) | week 0
  The SF-12 is a quality of life questionnaire. The scores range from 0 (worst conceivable QOL) to 100 (best conceivable QOL)
Short-form 12 questionnaire (SF-12) | week 7
  The SF-12 is a quality of life questionnaire. The scores range from 0 (worst conceivable QOL) to 100 (best conceivable QOL)
6 minute walking test | week 0
  walking distance
6 minute walking test | week 7
  walking distance
daily steps | week0
  the number of total walking steps per day which is measured by pedometer.
daily steps | week 7
  the number of total walking steps per day which is measured by pedometer.

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Huey Chen, PhD, Principal Investigator — Chang Gung University
Locations (1):
- Taoyuan General Hospital, Taoyuan District, Taiwan